CLINICAL TRIAL: NCT04232865
Title: Biop System's Safety and Performance in Increased Detection of High-grade Lesions of the Cervical Epithelium in Women Scheduled for Colposcopy
Brief Title: Biop System's Safety and Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BIOP Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP - 432
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bןםפ Sטדאקצ (Experimental): Biop Colposcopy procedure
  Interventions: Device: Biop System

INTERVENTIONS:
Device: Biop System — Stage 1 - Training:
  Up to 320 women in whom a complete procedure with the Biop System will be performed. Biopsies will be taken solely based on colposcopy examination. Enrolled participants will include at least 80 participants Histopathology identified with a high-grade lesion and at least 80 participants Histopathology identified as normal or with a low-grade lesion.
  Stage 2 - Validation:
  Up to 330 HIV negative women in whom a complete procedure with the Biop System will be performed.
  Validation stage will also include up to 165 HIV positive participants. All participants will be enrolled in up to 3 sites in South Africa.
  Other Names: Biop Colposcopy System

SUMMARY:
Biop system's safety and performance in increased detection of High-Grade lesions of the cervical epithelium in women scheduled for colposcopy

DETAILED DESCRIPTION:
Biop system's safety and performance in increased detection of high-grade lesions of the cervical epithelium in women scheduled for colposcopy.

This is a multi-center, prospective, open label, non-randomized study to train the Biop System's algorithm and evaluate the safety and performance of the Biop system in women undergoing cervical colposcopy.

ELIGIBILITY:
Inclusion Criteria:

* Female Age ≥ 22 years and ≤ 65.
* Referred for colposcopy, following abnormal cervical cytology;
* Participant provides signed informed consent

Exclusion Criteria:

* Currently pregnant (through six weeks postpartum) or nursing
* Currently menstruating
* Previous hysterectomy
* Currently has intrauterine device (IUD)
* Cervical biopsy or therapeutic procedure since the referral cervical cytology,
* Diagnosed with diseases that may influence the color of the tissue, e.g., hepatitis, polycythemia vera.
* Known human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS) (Applicable to training stage only)
* A known latex allergy
* Psychological instability, inappropriate attitude or motivation
* Cervical cytology tests within the prior seven days
* Use of vaginal medications within the last 48 h or photosensitizing agents within 72 h
* History of photosensitivity or other diseases affected by UV radiation,
* An observable and untreated gynecological infection.
* Previous history of CIN therapy

Ages: 22 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 320 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
SAE | through study completion, an average of 1 year
  The primary safety endpoint will be consisted of frequency and incidence of all Device Related Adverse Events (AE) and Serious Adverse Events (SAE).
Performance | through study completion, an average of 1 year
  Incremental True positive (TP) rate and Incremental False positive (FP) rate

IPD SHARING:
Plan to Share IPD: No